CLINICAL TRIAL: NCT03398746
Title: The LOOP Trial: A Study Comparing the Use of the LOOP Technique Versus Standard Incision and Drainage in the Treatment of Skin Abscesses in a Level I Emergency Department
Brief Title: The LOOP Trial in Treatment of Skin Abscesses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Regional Medical Center (Other)
Responsible Party: Principal Investigator, Jay Ladde, Associate Program Director, Orlando Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.005.01
Record Dates: First submitted 2018-01-03; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Abscess
Keywords: soft tissue infection; MRSA
MeSH Terms: conditions — Abscess; Soft Tissue Infections | interventions — LAMP assay; Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LOOP Technique (Experimental): Placement of subcutaneous loop drain
  Interventions: Procedure: LOOP Technique
- Incision and Drainage (Active Comparator): Standard Incision and Drainage Technique
  Interventions: Procedure: Standard incision and drainage

INTERVENTIONS:
Procedure: LOOP Technique — Placement of subcutaneous loop drain
  Arms: LOOP Technique
Procedure: Standard incision and drainage — Incise and drain with placement of packing
  Arms: Incision and Drainage

SUMMARY:
This prospective, randomized controlled trial enrolled a convenience sample of adults and children presenting to two Level 1 trauma centers over 12-months with subcutaneous skin abscesses necessitating drainage. Two methods of drainage were compared: 1) the LOOP technique or 2) standard packing technique.

DETAILED DESCRIPTION:
This prospective, randomized controlled trial enrolled a convenience sample of adults and children presenting to two Level 1 trauma centers over 12-months with subcutaneous skin abscesses necessitating drainage. Patients were excluded if the abscess was on the hand, foot, or face or if it required admission or operative intervention. Patients were followed over 10 days to determine the primary outcome of treatment failure defined by need for admission, IV antibiotics, or repeat drainage within 10-day follow-up. The secondary outcomes included ease of procedure, ease of care, pain after insertion and patient satisfaction using a 10-point numeric rating.

ELIGIBILITY:
Inclusion Criteria:

* Subcutaneous skin abscesses necessitating drainage

Exclusion Criteria:

* Abscess was on the hand, foot, or face
* Requiring admission or operative intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2009-01-22 (Actual); Primary Completion 2012-11-05 (Actual); Study Completion 2012-11-05 (Actual)

PRIMARY OUTCOMES:
Treatment Failure | 10 Days
  Need for admission, IV antibiotics, or repeat drainage within 10-day follow-up derived from descriptive nature

SECONDARY OUTCOMES:
Procedure Pain | At time of procedure
  Procedure Pain using Likert scale 1-10
Ease of procedure | At time of procedure
  Ease of procedure using Likert 1-10 scale
Ease of care | During 10 days
  Ease of care using 1-10 Likert scale
Pain on follow-up | 10 days
  Pain on follow-up using 1-10 Likert scale
Patient satisfaction | During 10 days
  Patient satisfaction using Patient derived Likert scale

REFERENCES:
- [Background] Ladde JG, Baker S, Rodgers CN, Papa L. The LOOP technique: a novel incision and drainage technique in the treatment of skin abscesses in a pediatric ED. Am J Emerg Med. 2015 Feb;33(2):271-6. doi: 10.1016/j.ajem.2014.10.014. Epub 2014 Oct 16. PMID 25435407
- [Derived] Ladde J, Baker S, Lilburn N, Wan M, Papa L. A Randomized Controlled Trial of Novel Loop Drainage Technique Versus Standard Incision and Drainage in the Treatment of Skin Abscesses. Acad Emerg Med. 2020 Dec;27(12):1229-1240. doi: 10.1111/acem.14106. Epub 2020 Oct 11. PMID 32770686
- See also: Link to PubMed Article — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=PubMed&dopt=Citation&list_uids=25435407